CLINICAL TRIAL: NCT04036318
Title: Evaluation of Presumptive Periodic Treatment (PPT) of Sexually Transmitted Infections (STIs) Among High-risk Populations Including Men Who Have Sex With Men, Female Sex Workers (FSW) and Mining Populations in Tanzania.
Brief Title: Evaluation of Presumptive Periodic Treatment (PPT) of Sexually Transmitted Infections (STIs)
Acronym: PPT
Status: Completed | Type: Observational
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Dr. Amani Shao, Research Scientist, National Institute for Medical Research, Tanzania
Other Study IDs: 16.02.PPT
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Sexually Transmitted Diseases, Bacterial; HIV Infections
Keywords: Sexually Transmitted Infections; Periodic Presumptive Treatment
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial; HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Anorectal swabs, Endocervical swabs and dry swabs from ulcerative lesions will be collected for the assessment of the bacterial sexually transmitted infections. In addition, swabs will be taken from urethral discharges in men. 5 milliliters of blood will be collected from each study participant assessment of viral infections such as HIV and viral hepatitis (HBV and HCV)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sexually transmitted infections (STI) are important causes of reproductive health morbidity and mortality, and have long been implicated as major co-factors in the sexual transmission of HIV. Both ulcerative and non-ulcerative STI have been found to be strongly associated with HIV in cross-sectional and prospective studies and hence STI prevention and care are important aspects of HIV prevention.

Periodic Presumptive Treatment of STIS (PPT) where risk populations are presumptively treated with a single dose of Azithromycin+Cefixime in regular intervals of 3 months has been shown to be effective in reducing STI prevalence at population level and has recently been integrated into the National STI guidelines of Tanzania. The USAID funded Sauti program will be one of the first to implement these new guidelines and roll out PPT in high risk populations in selected regions in Tanzania. This study will evaluate the impact of PPT as delivered by the Sauti program on prevalence of STIs in men who have sex with men and female sex workers in Dar es Salaam and Shinyanga respectively.

DETAILED DESCRIPTION:
This intervention linked study evaluates the impact of PPT on population level in FSW and MSM in Tanzania (Shinyanga and Dar es Salaam respectively). It is expected that PPT will reduce laboratory diagnosed STIs by 50% in the population after a roll out of 6 months.

This evaluation uses a cross-sectional venue-based sampling design. Three rounds of cross sectional data collection will be undertaken for MSM in Dar es Salaam and FSW in Shinyanga at three months intervals (baseline, 3 months and 6 months). The change in prevalence will be measured between baseline and 6 months assessments. The interim assessment will be used to refine the sample size. Study participants will be recruited in venues frequented by FSW (Shinyanga) and MSM (Dar es Salaam) in wards where Sauti operates. Respondents will be continuously sampled from all venues until sample size is reached. In each round of data collection, study participants will undergo physical examination, biological specimen collection, laboratory and HIV tests and a questionnaire.

STI prevalence in MSM and FSWs will be measured during each survey and laboratory-confirmed STI prevalence (gonorrhoea, chlamydia, syphilis) will be assessed.

Additionally, effect on STI prevalence in the bridge population will be measured by retrospective analysis of routine data for the prevalence of syndromic STIs among the mining population in Shinyanga, as collected in the context of the Sauti program mobile biomedical services (CBHTC+), which will visit the major mines in Shinyanga prior PPT implementation and after each survey. By the term major mines, we mean mines with large population of male mine workers (between 1000-2000 male mine workers) at higher risk of HIV rather than mines with modern mining infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give oral informed consent
* 18 years of age or older
* Is referred from the pre-selected recruitment venues and present and recruitment card.
* Sexually active in the last 6 months
* At least half of self-reported monthly income is generated through sex work (FSWs only)
* Men who engage in sexual relations with other men regardless of the motivation (MSMs only)

Exclusion Criteria:

* Not willing to give informed consent
* Not sexually active in the last 6 months
* State of intoxication from recreational drugs or alcohol use or other reasons which would prevent voluntary and informed consent to the study as judged by investigator
* Pregnant women - (determined through pregnancy screening questions used by Sauti)
* Does not have a study referral card

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to reach men who have sex with men (MSM) in Dar es Salaam region and female sex workers (FSWs) in Shinyanga region both of which are representative of the population in Tanzania.
  The study also is expected to have an effect on the bridging population in Shinyanga region. Bridge population in Shinyanga, are male mine workers who are considered to benefit from PPT provided to Female sex workers by Sauti program.
Sampling Method: Non-Probability Sample
Enrollment: 3022 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Reduction of prevalence of laboratory confirmed bacterial STIs | After six months of periodic presumptive treatment of STIs
  Reduction in prevalence of laboratory confirmed STIs (a combined measure of gonorrhea, chlamydia and Treponema pallidum) in men who have sex with men (MSMs) in Dar es Salaam and female sex workers (FSWs) in Shinyanga after six months of presumptive treatment of STIs (PPT).
Reduction of prevalence of syndromic STIs | After six months of periodic presumptive treatment of STIs among FSW in Shinyanga
  Syndromic STI prevalence (Genital ulcers disease (GUD), Anorectal Syndrome (ARS), Urethral Discharge Syndrome (UDS), Painful scrotal swelling (PSS)) among male clients of FSW in Shinyanga mines (bridge population) after six months of availability of PPT to FSWs. initiation.

SECONDARY OUTCOMES:
Associations between demographic, socio-economic, behavioral and biological risk factors, STI prevalence and PPT impact. | After six months of periodic presumptive treatment of STIs among FSW in Shinyanga
  The association will determined by using the logistic regression
Changes in sexual risk taking behaviors while receiving PPT | Six months
  Changes in sexual risk behaviors will be determined by comparing the baseline prevalence and prevalence after six months of PPT
Prevalence of cervical cancer lesions | Six months
  The prevalence of cervical cancer lesions, will be assessed through Visual Inspection with Acetic Acid (VIA), among the FSW in the study.
Prevalence of Human Papilloma Virus (HPV), HIV, Hepatitis B and C | Six months
  The prevalence of Human Papilloma Virus (HPV), HIV, Hepatitis B and C will be assessed from the bio-specimens of serum and genital swabs collected during the surveys

CONTACTS AND LOCATIONS:
Overall Officials: Amani Shao, MD; MPH; PhD, Principal Investigator — National Institute for Medical Research
Locations (2):
- Tanzania (2):
  - Shinyanga Region, Shinyanga, Kahama
  - Dar es Salaam region, Dar es Salaam, Temeke

IPD SHARING:
Plan to Share IPD: Yes
As part of the open data policy, all data emanating from this study will be shared with other researchers
Supporting Information: Study Protocol, ICF
Time Frame: The IPD will be shared during the study closure
Access Criteria: Will be determined by the funder and sponsor